CLINICAL TRIAL: NCT05386251
Title: Effectiveness of a Digital Strategy-based Educational Skills Group for Secondary Students With Organization and Academic Motivation Challenges
Acronym: STAND-G
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Margaret Sibley, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00003308
Record Dates: First submitted 2021-09-24; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: ADHD
Keywords: ADHD; Behavioral Intervention; Telehealth
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Students are randomized in a 1:1 allocation ratio to the active treatment of the control group. Participants will be randomized to the strategies or peer support groups using a stratified randomization procedure that randomizes within grade level (i.e., middle school or high school). After 20 students are randomized to a group, the group will be scheduled to begin.
Who Masked: Participant, Outcomes Assessor
Masking Description: The same providers will deliver both treatment arms and so it will be difficult to fully mask the providers to which group is active (based on their natures). However, participants will be told that both groups are active and outcomes assessors will not be informed about group membership.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Parent Training/Organization Skills Training (Experimental): Parents will receive 8 weeks of a 90 minute behavioral parent training protocol that focuses on supporting academic and behavioral success in adolescents with ADHD. Teens will receive a simultaneous 8 weeks of a 90 minute organization skills training group. Both groups will be delivered via telehealth.
  Interventions: Behavioral: BPT/OST
- Peer support (Sham Comparator): Parents and teens will each participate in 8 weeks of a 90 minute peer support group focused on exchange of shared experience and group problem-solving difficulties. Both groups will be delivered via telehealth.
  Interventions: Behavioral: Peer Support

INTERVENTIONS:
Behavioral: BPT/OST — See Arm description.
  Other Names: STAND-Group
  Arms: Behavioral Parent Training/Organization Skills Training
Behavioral: Peer Support — See Arm description
  Arms: Peer support

SUMMARY:
The purpose of this study is to test the effectiveness of a telehealth-delivered skills training versus active control group for middle and high school students with ADHD symptoms. Both programs will be delivered digitally (via Zoom).

Investigators will measure student functioning at baseline, post-group, and three-month follow-up. The primary outcomes are ADHD symptoms, student grade point average, and attendance as reported in the gradebook. Secondary outcomes include parent academic support, autonomy, academic motivation, and organization skills. Participant satisfaction with the group will be measured post-group. Group attendance and homework completion will also be measured.

DETAILED DESCRIPTION:
120 middle and high school students with elevated ADHD symptoms will be recruited for this study, which will take place over the course of the 2021-2022 academic year. The recruitment strategy will be to distribute information about the study opportunity to educator email lists in South Florida (see appended email template). Educators will be instructed to share information about the study to the parents of students who perceive to experience ADHD symptoms in their schools, regardless of special education status or documentation of a disability.

Students who enroll will be randomly assigned to either receive the STAND-G strategy-based group or a peer-support-based, active control group. Investigators will blind participants and their parents to which group is the active treatment by informing parents and students that participant will be randomly assigned to one of two groups to help improve school difficulties in youth. The two groups will be of equal duration, both will be led by the same instructors; and will differ only in content (teaching strategies vs. facilitating peer support and problem-solving conversations).

Students (and their parents) will complete assessments at baseline, post-group, and three months post-group. School records will be obtained for all time points.

ELIGIBILITY:
Inclusion Criteria:

Students will be required to,

* be in the sixth through twelfth grade,
* have elevated ADHD symptoms
* documented impairment according to the SNAP
* documented impairment according to Impairment Rating Scale.
* Students must be 17.5 or younger at the time of enrollment to ensure that they are still under 18 at the expected completion of the study.

Parents of eligible students will also participate.

Exclusion Criteria:

Students may not be,

* in a self-contained special education classroom,
* possess intellectual disability
* be non-English speaking
* be older than 18 years old at time of enrollment

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-05-18 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
ADHD Symptoms | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  Parent and Self Ratings on the SNAP Rating Scale
Academic Impairment: Grade Point Average | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  Official School Records
Academic Impairment: School Attendance | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  Official School Records

SECONDARY OUTCOMES:
Academic Motivation | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  Expectancy-Value Questionnaire -Self Version
Academic Motivation | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  Change Ruler -Self Version
Executive Functions | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  BRIEF Rating Scale -Parent Version
Organization, Time Management, and Planning | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  Adolescent Academic Problems Checklist-Parent and Self Version will be used to measure organization, time management and planning
Parent Academic Involvement | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  Parent Academic Management Scale - Parent Version
Academic Impairment Rating Scale | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  Impairment Rating Scale - Parent Version
Parent-Teen Conflict | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  Conflict Behavior Questionnaire-20 - Parent, Self Version
Goal Setting | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  Goal Setting Questionnaire- Parent and Self
Parent Autonomy Support | Change from Baseline through 3 months after Post-Treatment, an average of 6 months
  Parent Promotion of Volitional Functioning- Self Report

OTHER OUTCOMES:
Treatment Satisfaction | At Post-treatment, approximately 8 weeks after initial group session
  Parent and Self Report Satisfaction Survey
Treatment Fidelity | Through Treatment Completion, an average of 8 weeks
  Blinded Observers will observe to code for fidelity
Treatment Barriers | At Post-treatment, approximately 8 weeks after initial group session
  Parent an Self Reported Barriers Survey
Treatment Credibility | At Post-treatment, approximately 8 weeks after initial group session
  Client Credibility Questionnaire-Parent and Self
Video Conferencing Feasibility | At Post-treatment, approximately 8 weeks after initial group session
  Video-Conferencing Questionnaire-Parent and Self
Treatment Attendance | Through study completion, an average of 8 weeks, at each Session of Treatment
  Group records
Treatment Homework Completion | Through study completion, an average of 8 weeks, at each Session of Treatment
  Group records

IPD SHARING:
Plan to Share IPD: Yes
We will submit data from this trial to the OSF data repository upon completion of the trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within six months of the completion of the trial